CLINICAL TRIAL: NCT02013362
Title: Phase I/II Clinical Study of Pralatrexate in Japanese Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mundipharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-JP1
Record Dates: First submitted 2013-12-04; First posted 2013-12-17 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pralatrexate injection (Experimental): Dietary Supplement: Vitamin B12, Folic Acid
  Interventions: Drug: Pralatrexate injection; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate injection
Dietary Supplement: Vitamin B12
Dietary Supplement: Folic Acid

SUMMARY:
Phase I portion:

To evaluate the safety and tolerability of pralatrexate with concurrent vitamin B12 and folic acid supplementation in Japanese patients with relapsed or refractory PTCL and to determine the recommended dosage. Also, to evaluate pharmacokinetics.

Phase II portion:

To evaluate the efficacy, safety, and pharmacokinetics of the recommended dosage regimen determined in the phase I portion. The primary efficacy endpoint shall be objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients at least 20 years of age.
* Patients histologically diagnosed with peripheral T-cell lymphoma by pathological diagnosis of biopsied lesion.
* Relapsed or refractory patients with a treatment history of at least one regimen.
* Patients with an enlarged lymph node or extranodal mass lesion clearly measurable in two perpendicular directions and greater than 1.5 cm in maximum diameter on computed tomography performed.
* Patients expected to survive for at least 3 months.
* ECOG PS 0-2.
* Patients with adequate hemopoietic efficacy, liver and kidney function.
* Patients from whom written consent has been obtained prior to study initiation.

Exclusion Criteria:

* Patients who received a chemotherapy agent or a high dose of a systemic adrenocorticosteroid within 21 days prior to initial administration of the study drug.
* Patients who received radiation therapy, phototherapy, or electron beam therapy within 21 days prior to initial administration of the study drug.
* Patients who received another study drug within 28 days prior to initial administration of the study drug.
* Patients who received antibody therapy within 100 days prior to initial administration of the study drug.
* Patients with a history of allogeneic hematopoietic stem cell transplantation. Or patients with a history of autologous hematopoietic stem cell transplantation within 100 days prior to initial administration of the study drug.
* Patients with cerebral metastasis or central nervous system lesion or a past history.
* Patients with active multiple primary cancer. Or patients with a history of a malignant neoplasm other than peripheral T-cell lymphoma within the past 5 years.
* Patients with severe cardiovascular disease.
* Patients positive for HBs antigen, HCV antibody or HIV antibody on immunological investigation. Or patients positive for either HBc antibody or HBs antibody, and showing DNA more than sensitivity in HBV-DNA assay.
* Patients positive for CMV antigen on immunological investigation.
* Patients with infectious disease requiring treatment consisting of intravenous administration of antibacterial agent, fungicide, or antiviral drug.
* Patients with interstitial pneumonia or pulmonary fibrosis, or patients judged to have insufficient pulmonary function.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) per independent central review committee | From screening period until first documented disease progression or treatment discontinuation from any cause, whichever came first. Duration is approximately 3 years.
  The ORR is defined as the proportion of patients with complete response (CR) and partial response (PR). Response will be determined according to International Workshop Criteria (IWC). Assessments will be done at week 7 (end of Cycle 1), subsequently every 14 weeks (end of odd-numbered cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD,PhD, Principal Investigator — National Cancer Center Hospital
Locations (3):
- Japan (3):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital, Chūō, Tokyo
  - Okayama University Hospital, Okayama

REFERENCES:
- [Derived] Maruyama D, Nagai H, Maeda Y, Nakane T, Shimoyama T, Nakazato T, Sakai R, Ishikawa T, Izutsu K, Ueda R, Tobinai K. Phase I/II study of pralatrexate in Japanese patients with relapsed or refractory peripheral T-cell lymphoma. Cancer Sci. 2017 Oct;108(10):2061-2068. doi: 10.1111/cas.13340. Epub 2017 Sep 4. PMID 28771889